CLINICAL TRIAL: NCT03583333
Title: A Multi-national Phase 3, Randomized, Double-Blind, Active Comparator-Controlled Clinical Trial to Study the Safety, Tolerability, and Efficacy of Imipenem/Cilastatin/Relebactam (MK-7655A) Versus Piperacillin/Tazobactam in Subjects With Hospital-Acquired Bacterial Pneumonia or Ventilator-Associated Bacterial Pneumonia
Brief Title: Imipenem/Cilastatin/Relebactam (MK-7655A) Versus Piperacillin/Tazobactam in Participants With Hospital-Acquired or Ventilator-Associated Bacterial Pneumonia (MK-7655A-016)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7655A-016; MK-7655A-016 (Other: MSD Protocol Number); PHRR190814-002177 (Registry Identifier: PHRR); 2018-003202-82 (EudraCT Number)
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Hospital-Acquired Bacterial Pneumonia; Ventilator-Associated Bacterial Pneumonia
MeSH Terms: interventions — Linezolid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IMI/REL FDC (Experimental): Imipenem/cilastatin/relebactam (IMI/REL) administered intravenously (IV) as a fixed-dose combination (FDC) at a dosage of 500 mg IMI/250 mg REL, once every 6 hours for a minimum 7 days, up to 14 days. At the start of IMI/REL treatment, participants will be treated empirically with 600 mg open-label linezolid administered IV every 12 hours until methicillin-resistant Staphylococcus aureus (MRSA) is ruled out. Participants with confirmed MRSA infection will continue to receive 600 mg linezolid every 12 hours for a minimum of 7 days, up to 14 days total.
  Interventions: Drug: IMI/REL FDC; Drug: Linezolid
- PIP/TAZ FDC (Active Comparator): Piperacillin/tazobactam (PIP/TAZ ) administered IV as a FDC at a dosage of 4000 mg PIP/500 mg TAZ once every 6 hours for a minimum 7 days, up to 14 days. At the start of PIP/TAZ treatment, participants will be treated empirically with 600 mg open-label linezolid administered IV every 12 hours until methicillin-resistant Staphylococcus aureus (MRSA) is ruled out. Participants with confirmed MRSA infection will continue to receive 600 mg linezolid every 12 hours for a minimum of 7 days, up to 14 days total.
  Interventions: Drug: PIP/TAZ FDC; Drug: Linezolid

INTERVENTIONS:
Drug: IMI/REL FDC — 500 mg Imipenem, 500 mg Cilastatin and 250 mg Relebactam powder FDC provided in a single vial
  Other Names: MK-7655A
  Arms: IMI/REL FDC
Drug: PIP/TAZ FDC — 4000 mg Piperacillin and 500 mg Tazobactam powder FDC provided in a single vial
  Arms: PIP/TAZ FDC
Drug: Linezolid — Open-label 600 mg Linezolid

SUMMARY:
This study will evaluate the efficacy and safety of a FDC of imipenem/cilastatin (IMI) and relebactam (REL) [IMI/REL, MK-7655A] compared to piperacillin/tazobactam (PIP/TAZ) in the treatment of adults diagnosed with Hospital-Acquired Bacterial Pneumonia (HABP) or Ventilator-Associated Bacterial Pneumonia (VABP). The primary hypothesis is that IMI/REL is non-inferior to PIP/TAZ as measured by the incidence rate of all-cause mortality through Day 28 post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Requires treatment with IV antibiotic therapy for HABP or VABP
* Fulfills clinical and radiographic criteria within 48 hours prior to randomization, with onset of criteria occurring after more than 2 days of hospitalization or within 7 days after discharge from a hospital for HABP; or at least 2 days after mechanical ventilation (for VABP)
* Has an adequate baseline (at or within 2 days of screening) lower respiratory tract specimen obtained for Gram stain and culture
* Has an infection known or thought to be, in the opinion of the investigator, caused by microorganisms susceptible to the IV study therapy
* Agrees to allow any bacterial isolates obtained from protocol-required specimens related to the current infection to be provided to the Central Microbiology Reference Laboratory for study-related microbiological testing and long-term storage
* Males agree to use contraception as detailed in protocol from the time of providing informed consent through completion of the study and refrain from donating sperm during this period
* Females are not pregnant, not breastfeeding, and are either: a.) Not a woman of childbearing potential (WOCBP) OR b.) A WOCBP who agrees to follow the contraceptive guidance from the time of providing informed consent through completion of the study
* If a penicillin skin test is required by local clinical practice, the participant must have a negative skin test result for allergy to penicillin

Exclusion Criteria:

* Has a baseline lower respiratory tract specimen Gram stain that shows the presence of Gram-positive cocci only
* Has confirmed or suspected community-acquired bacterial pneumonia (CABP)
* Has confirmed or suspected pneumonia caused by Mycoplasma, Chlamydia, or Legionella, or of viral, fungal, or parasitic etiology
* Has HABP/VABP caused by an obstructive process, including lung cancer (or other malignancy metastatic to the lungs resulting in pulmonary obstruction) or other known obstruction
* Has a carcinoid tumor or carcinoid syndrome
* Has active immunosuppression
* Is expected to die during the 7- to 14-day treatment period, despite adequate antibiotic therapy
* Has a concurrent condition or infection that, in the investigator's judgment, would preclude evaluation of therapeutic response
* Has a history of serious allergy, hypersensitivity, or any serious reaction to any β-lactams or β-lactamase inhibitors
* Has a history of a seizure disorder which has required ongoing treatment with anticonvulsive therapy or prior treatment with anti-convulsive therapy within the last 3 years
* Is currently undergoing hemodialysis or peritoneal dialysis
* A WOCBP who has a positive urine pregnancy test at screening
* Has received effective antibacterial drug therapy with known coverage of pathogens that cause HABP/VABP for a continuous duration of more than 48 hours during the previous 72 hours
* Is anticipated to be treated with any of the prohibited medications during the course of study therapy
* Is currently participating in, or has participated in, any other clinical study involving the administration of investigational or experimental medication (not licensed by regulatory agencies) at the time of the presentation or during the previous 90 days prior to screening or is anticipated to participate in such a clinical study during the course of this trial
* Has previously participated in this study at any time

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (68):
- Brazil (2):
  - Santa Casa de Misericordia de Belo Horizonte ( Site 0300), Belo Horizonte, Minas Gerais
  - Hospital de Base de Sao Jose de Rio Preto ( Site 0301), Sao Jose Do Rio Preto - SP, São Paulo
- China (45):
  - Beijing Chaoyang Hospital ( Site 0126), Beijing, Beijing Municipality
  - Peking University First Hospital ( Site 0131), Beijing, Beijing Municipality
  - Aero Space center hospital ( Site 0118), Beijing, Beijing Municipality
  - The Seventh Medical Center of PLA General Hospital-Intensive medicine ( Site 0157), Beijing, Beijing Municipality
  - Peking University Third Hospital ( Site 0115), Beijing, Beijing Municipality
  - Beijing Hospital ( Site 0127), Beijing, Beijing Municipality
  - The First Affiliated Hospital Of Fujian Medical University-Respiratory ( Site 0136), Fuzhou, Fujian
  - Zhongshan Hospital Affiliated to Xiamen University ( Site 0133), Xiamen, Fujian
  - Zhangzhou Municipal Hospital of Fujian Province-Neurosurgery Department ( Site 0150), Zhangzhou, Fujian
  - The First Affiliated Hospital ( Site 0100), Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University ( Site 0123), Guangzhou, Guangdong
  - Guangzhou First People's Hospital ( Site 0101), Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University ( Site 0148), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital ( Site 0120), Guangzhou, Guangdong
  - Huizhou Municipal Central Hospital ( Site 0140), Huizhou, Guangdong
  - Shenzhen People s Hospital ( Site 0134), Shenzhen, Guangdong
  - The first people s hospital of Nanning ( Site 0138), Nanning, Guangxi
  - The first people s hospital of Nanning ( Site 0141), Nanning, Guangxi
  - Hainan General Hospital ( Site 0106), Haikou, Hainan
  - The First Affiliated Hospital of Zhengzhou University ( Site 0121), Zhengzhou, Henan
  - Shiyan City People's Hospital-Neurosurgery ( Site 0155), Shiyan, Hubei
  - Changsha Central Hospital ( Site 0119), Changsha, Hunan
  - Hunan Provincial People Hospital ( Site 0122), Changsha, Hunan
  - The First People's Hospital of Changzhou ( Site 0139), Changzhou, Jiangsu
  - First Huai'an Hospital Affiliated to Nanjing Medical University-Neurosurgery Department ( Site 0153), Huai'an, Jiangsu
  - First Hospital Affiliated to Suzhou University ( Site 0111), Suzhou, Jiangsu
  - Wuxi People's Hospital ( Site 0124), Wuxi, Jiangsu
  - Affiliated Hospital of Jiangsu University ( Site 0147), Zhenjiang, Jiangsu
  - Jiangxi Provincial People's Hospital ( Site 0129), Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University ( Site 0132), Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University-Neurosurgery Department ( Site 0151), Nanchang, Jiangxi
  - The First Affiliated Hospital of China Medical University ( Site 0116), Shenyang, Liaoning
  - General Hospital of Ningxia Medical University ( Site 0135), Yinchuan, Ningxia
  - People's Hospital of Liaocheng City-Neurology ( Site 0154), Liaocheng, Shandong
  - Ruijin Hospital Shanghai Jiao Tong University School of Medicine ( Site 0104), Shanghai, Shanghai Municipality
  - Huadong Hospital Affiliated Fudan University ( Site 0103), Shanghai, Shanghai Municipality
  - Huashan Hospital of Fudan University ( Site 0105), Shanghai, Shanghai Municipality
  - Shanghai General Hospital ( Site 0125), Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital ( Site 0108), Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital ( Site 0113), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital.Zhejiang University ( Site 0102), Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital School of Medicine Zhejiang University ( Site 0110), Hangzhou, Zhejiang
  - People s Hospital of Lishui City ( Site 0137), Lishui, Zhejiang
  - Ningbo First Hospital-neurosurgery ( Site 0152), Ningbo, Zhejiang
  - The 2nd Affiliated Hospital of Wenzhou Medical University ( Site 0130), Wenzhou, Zhejiang
- France (4):
  - Hopital Roger Salengro du Lille ( Site 0601), Lille, Nord
  - CHU de Nantes - Hotel Dieu ( Site 0600), Nantes, Pays de la Loire Region
  - Hospices Civils de Lyon ( Site 0603), Pierre-Bénite, Rhone
  - Hopital Bicetre ( Site 0605), Le Kremlin-Bicêtre, Val-de-Marne
- Mexico (2):
  - Hospital Civil de Guadalajara Fray Antonio Alcalde ( Site 0800), Guadalajara, Jalisco
  - Hospital Civil Nuevo de Guadalajara Dr. Juan I. Menchaca ( Site 0804), Guadalajara, Jalisco
- Philippines (3):
  - Mary Johnston Hospital ( Site 0901), Metro Manila, National Capital Region
  - Lung Center of the Philippines ( Site 0903), Quezon City, National Capital Region
  - West Visayas State University Medical Center ( Site 0900), Iloilo City
- Romania (2):
  - Spitalul Clinic Judetean de Urgenta Pius Branzeu ( Site 1103), Timișoara, Timiș County
  - Spitalul Clinic de Urgenta Bagdasar-Arseni ( Site 1101), Bucharest
- Russia (5):
  - First City Clinical Hospital n.a. E.E.Volosevich ( Site 1016), Arkhangelsk, Arkhangelskaya oblast
  - City Hospital #2 Severodvinsk ( Site 1017), Severodvinsk, Arkhangelskaya oblast
  - Research Institute of Emergency Medicine n.a. I.I.Dzhanelidze ( Site 1011), Saint Petersburg, Sankt-Peterburg
  - Clinical Hospital #122 L.G. Sokolova FMBA ( Site 1015), Saint Petersburg, Sankt-Peterburg
  - City Hospital #26 ( Site 1002), Saint Petersburg, Sankt-Peterburg
- Ukraine (5):
  - ME Dnipropetrovsk Clinical Joinder of Emergency Care of DRC ( Site 1304), Dnipro, Dnipropetrovsk Oblast
  - Ivano-Frankivsk regional clinical hospital ( Site 1301), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - City Clinical Hospital No13 of Kharkiv City Council ( Site 1303), Kharkiv, Kharkivs’ka Oblast’
  - Kiyv city municipal hospital 17 ( Site 1300), Kiev, Kyivska Oblast
  - Reg. Clin. Hospital ( Site 1306), Poltava, Poltava Oblast

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Li J, Wei F, Xiang P, Tang Z, Ding L, Chen LF, Losada M, Iamboliyska Z, Sun F, Zhu M, Guo X, Du X, Chen C, Bruno C, Koseoglu S, Young K, Zhou M, Qu J. A phase III, randomized, controlled noninferiority trial to study the efficacy and safety of imipenem/cilastatin/relebactam (IMI/REL) vs piperacillin/tazobactam (PIP/TAZ) in patients with hospital-acquired bacterial pneumonia (HABP) or ventilator-associated bacterial pneumonia (VABP). Int J Infect Dis. 2025 Apr;153:107357. doi: 10.1016/j.ijid.2024.107357. Epub 2024 Dec 12. PMID 39674398

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 54 centers in 8 countries.
Pre-assignment Details: Participants were randomized 1:1 to receive either FDC of imipenem/cilastatin (IMI) and relebactam (REL) [IMI/REL, MK-7655A], or piperacillin/tazobactam (PIP/TAZ).
Groups:
- IMI/REL FDC: Imipenem/cilastatin/relebactam (IMI/REL) was administered intravenously (IV) as a fixed-dose combination (FDC) at a dosage of 500 mg IMI/250 mg REL, once every 6 hours for a minimum 7 days, up to 14 days. At the start of IMI/REL treatment, participants were treated empirically with 600 mg open-label linezolid administered IV every 12 hours until methicillin-resistant Staphylococcus aureus (MRSA) was ruled out. Participants with confirmed MRSA infection continued to receive 600 mg linezolid every 12 hours for a minimum of 7 days, up to 14 days total.
- PIP/TAZ FDC: Piperacillin/tazobactam (PIP/TAZ) was administered IV as a FDC at a dosage of 4000 mg PIP/500 mg TAZ once every 6 hours for a minimum 7 days, up to 14 days. At the start of PIP/TAZ treatment, participants were treated empirically with 600 mg open-label linezolid administered IV every 12 hours until methicillin-resistant Staphylococcus aureus (MRSA) is ruled out. Participants with confirmed MRSA infection continued to receive 600 mg linezolid every 12 hours for a minimum of 7 days, up to 14 days total.
Period: Overall Study
Arm/Group | IMI/REL FDC | PIP/TAZ FDC
Started | 138 | 136
Treated | 134 | 136
Completed | 90 | 106
Not Completed | 48 | 30
Not completed — Participant Conducted Day 28 Visit Prior to the Required Time Window | 8 | 6
Not completed — Withdrawal by Parent/Guardian | 16 | 10
Not completed — Withdrawal by Subject | 9 | 5
Not completed — Physician Decision | 3 | 2
Not completed — Death | 12 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IMI/REL FDC | PIP/TAZ FDC | Total
Number analyzed (Participants) | 138 | 136 | 274
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.9 (15.1) | 59.2 (14.7) | 57.5 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 36 | 73
  Male | 101 | 100 | 201
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 12
  Not Hispanic or Latino | 134 | 128 | 262
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 110 | 102 | 212
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 27 | 33 | 60
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Randomization strata: Pneumonia type at baseline [Count of Participants; unit: Participants] — Participants were stratified by the following two pneumonia types at baseline: Non-ventilated hospital acquired bacterial pneumonia (HABP) and ventilated HABP/ventilator associated bacterial pneumonia (VABP).
  Participants
    Non-ventilated HABP | 74 | 80 | 154
    Ventilated HABP/VABP | 64 | 56 | 120
Randomization strata: Acute Physiology and Chronic Health Evaluation (APACHE) II score at baseline [Count of Participants; unit: Participants] — APACHE score is a severity-of-disease classification system that is calculated from a participants age and 12 routine physiological measurements. Total scores are computed based on several measurements and range from 0 to 71 with higher scores corresponding to more severe disease and a higher risk of death. Participants were stratified by APACHE II score at baseline <15 vs. >15
  Participants
    APACHE II Score <15 | 65 | 61 | 126
    APACHE II Score ≥15 | 73 | 75 | 148

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With All-cause Mortality Through Day 28 in the Modified Intent to Treat (MITT) Population
Description: For each participant, survival status was assessed at Day 28 post-randomization and recorded on the electronic Case Report Form. The percentage of participants with all-cause mortality through Day 28 in the MITT population is presented.
Time Frame: Up to approximately 28 days
Population: The MITT population consisting of all randomized participants who received at least 1 dose of IV study therapy and did not have the presence of positive cocci only on baseline Gram stain were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | IMI/REL FDC | PIP/TAZ FDC
Number analyzed (Participants) | 134 | 136
Percentage of Participants | 11.2 | 5.9
Statistical Analysis 1: Comparison: IMI/REL FDC vs PIP/TAZ FDC; Test type: Non-Inferiority — Non-inferiority margin for the difference in mortality (IMI/REL minus PIP/TAZ) was 12.5%; p = 0.024, Miettinen & Nurminen method; Adjusted difference in percentage = 5.2, 95% CI 2-sided [-1.5 to 12.4] — Adjusted differences and the 95% confidence intervals (CIs) are based on Miettinen & Nurminen method stratified by randomization stratum
Statistical Analysis 2: Comparison: IMI/REL FDC vs PIP/TAZ FDC; Test type: Superiority; p = 0.938, Miettinen & Nurminen; Adjusted differences and the 95% CIs are based on Miettinen & Nurminen method stratified by randomization stratum; Adjusted difference in percentage = 5.2, 95% CI 2-sided [-1.5 to 12.4]

2. Secondary Outcome: Percentage of Participants Achieving a Favorable Clinical Response at Early Follow-up (EFU) Visit in the MITT Population
Description: Clinical response was defined as "Sustained cure" (All pretherapy signs and symptoms of the index infection have resolved or returned to preinfection status with no evidence of resurgence AND no additional antibiotic therapy was required for the index infection) or "Cure" (All pretherapy signs and symptoms of the index infection have resolved or returned to preinfection status AND no additional antibiotic therapy was required for the index infection). The percentage of participants achieving a favorable clinical response at EFU visit in the MITT population is presented.
Time Frame: Up to approximately 27 days
Population: MITT population consisting of all randomized participants who received at least 1 dose of IV study therapy and did not have the presence of positive cocci only on baseline Gram stain.
Measure: Number; unit: Percentage of Participants
Arm/Group | IMI/REL FDC | PIP/TAZ FDC
Number analyzed (Participants) | 134 | 136
Percentage of Participants | 50.7 | 47.8
Statistical Analysis 1: Comparison: IMI/REL FDC vs PIP/TAZ FDC; Test type: Other; Adjusted difference in percentage = 3.1, 95% CI 2-sided [-8.7 to 14.9] — Adjusted differences and the 95% CIs are based on Miettinen & Nurminen method stratified by randomization stratum

3. Secondary Outcome: Percentage of Participants Achieving a Favorable Clinical Response at EFU Visit in the Clinically Evaluable (CE) Population
Description: Clinical response was defined as "Sustained cure" (All pretherapy signs and symptoms of the index infection have resolved or returned to preinfection status with no evidence of resurgence) AND no additional antibiotic therapy was required for the index infection or "Cure" (All pretherapy signs and symptoms of the index infection have resolved or returned to preinfection status) AND no additional antibiotic therapy was required for the index infection. The percentage of participants achieving a favorable clinical response at EFU visit in the CE population is presented.
Time Frame: Up to approximately 27 days
Population: MITT population consisting of all randomized participants who received at least 1 dose of IV study therapy and did not have the presence of positive cocci only on baseline Gram stain. The CE population was a subset of the MITT population who also met important diagnostic criteria for entry into the study, had no significant deviation from the protocol and received the minimum duration of IV study therapy. Only participants with non-missing/non-indeterminate response were assessed at EFU visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | IMI/REL FDC | PIP/TAZ FDC
Number analyzed (Participants) | 79 | 82
Percentage of Participants | 64.6 | 62.2
Statistical Analysis 1: Comparison: IMI/REL FDC vs PIP/TAZ FDC; Test type: Other; Adjusted difference in percentage = 2.2, 95% CI 2-sided [-12.4 to 16.8] — Adjusted difference and the 95% CIs are based on Miettinen & Nurminen method stratified by randomization stratum

4. Secondary Outcome: Percentage of Participants Achieving a Favorable Clinical Response at End of Therapy (EOT) Visit in the MITT Population
Description: Clinical response was defined as "Improved" (The majority of pre-therapy signs and symptoms of the index infection have improved or resolved or returned to "pre-infection status" AND no additional antibiotic therapy was required) or "Cure" (All pretherapy signs and symptoms of the index infection have resolved or returned to preinfection status AND no additional antibiotic therapy was required for the index infection). The percentage of participants achieving a favorable clinical response at EOT visit in the MITT population is presented.
Time Frame: Up to approximately 14 days
Population: MITT population consisting of all randomized participants who received at least 1 dose of IV study therapy and did not have the presence of positive cocci only on baseline Gram stain were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | IMI/REL FDC | PIP/TAZ FDC
Number analyzed (Participants) | 134 | 136
Percentage of Participants | 71.6 | 68.4
Statistical Analysis 1: Comparison: IMI/REL FDC vs PIP/TAZ FDC; Test type: Other; Adjusted difference in percentage = 3.4, 95% CI 2-sided [-7.6 to 14.3] — Adjusted difference and the 95% CIs are based on Miettinen & Nurminen method stratified by randomization stratum

5. Secondary Outcome: Percentage of Participants Achieving a Favorable Clinical Response at EOT Visit in the Clinically Evaluable (CE) Population
Description: Clinical response was defined as "Improved" (The majority of pre-therapy signs and symptoms of the index infection have improved or resolved or returned to "pre-infection status" AND no additional antibiotic therapy is required) or "Cure" (All pretherapy signs and symptoms of the index infection have resolved or returned to preinfection status) AND no additional antibiotic therapy is required for the index infection. The percentage of participants achieving a favorable clinical response at End of Treatment (EOT) visit in the CE population is presented.
Time Frame: Up to approximately 14 days
Population: MITT population consisting of all randomized participants who received at least 1 dose of IV study therapy and did not have the presence of positive cocci only on baseline Gram stain. The CE population was a subset of the MITT population who also met important diagnostic criteria for entry into the study, had no significant deviation from the protocol and received the minimum duration of IV study therapy. Only participants with non-missing/non-indeterminate response were assessed at EOT visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | IMI/REL FDC | PIP/TAZ FDC
Number analyzed (Participants) | 106 | 96
Percentage of Participants | 77.4 | 82.3
Statistical Analysis 1: Comparison: IMI/REL FDC vs PIP/TAZ FDC; Test type: Other; Adjusted difference in percentage = -4.7, 95% CI 2-sided [-15.8 to 6.6] — Adjusted difference and the 95% CIs are based on Miettinen & Nurminen method stratified by randomization stratum

6. Secondary Outcome: Percentage of Participants Achieving a Favorable Microbiological Response at EOT Visit in Microbiological Modified Intent-To-Treat Population (mMITT) Population
Description: Favorable overall microbiological response rates were defined as "eradication" (A lower respiratory tract culture taken at the EOT visit showed eradication of the pathogen found at study entry) OR "presumed eradication" (No specimen taken because participant was deemed clinically cured or improved) of the baseline pathogen. The percentage of participants achieving a favorable microbiological response at EOT visit in the mMITT population is presented.
Time Frame: Up to approximately 14 days
Population: The MITT population consisted of all randomized participants who received at least 1 dose of IV study therapy and did not have the presence of positive cocci. The microbiological modified intention-to-treat (mMITT) population was a subset of the MITT population that possessed a baseline bacterial pathogen isolated from a lower respiratory tract (LRT) specimen that was identified as the cause of HABP/VABP and against which IMI/REL has been shown to have antibacterial activity.
Measure: Number; unit: Percentage of Participants
Arm/Group | IMI/REL FDC | PIP/TAZ FDC
Number analyzed (Participants) | 80 | 73
Percentage of Participants | 57.5 | 60.3
Statistical Analysis 1: Comparison: IMI/REL FDC vs PIP/TAZ FDC; Test type: Other; Adjusted difference in percentage = -2.4, 95% CI 2-sided [-17.8 to 13.1] — Adjusted differences and the 95% CIs are based on Miettinen & Nurminen method stratified by randomization stratum

7. Secondary Outcome: Percentage of Participants Achieving a Favorable Microbiological Response at EFU Visit in Microbiological-evaluable (ME) Population.
Description: A favorable by-pathogen microbiological response at EFU visit required "eradication" (A lower respiratory tract culture taken at the EFU visit showed eradication of the pathogen found at study entry) or "presumed eradication" (No specimen taken because participant was deemed clinically cured or improved) of the baseline pathogen. The percentage of participants achieving a favorable microbiological response at EFU visit in the ME population is presented.
Time Frame: Up to approximately 27 days
Population: All randomized participants receiving ≥1 dose of IV study therapy without presence of positive cocci (MITT); who met important diagnostic criteria for study with no significant protocol deviation and received minimum duration of IV study therapy (CE); had a baseline bacterial pathogen cause of HABP/VABP against which IMI/REL has antibacterial activity and results from a lower respiratory tract culture obtained at indicated time point (ME); and had non-missing/non-indeterminate response at EFU.
Measure: Number; unit: Percentage of Participants
Arm/Group | IMI/REL FDC | PIP/TAZ FDC
Number analyzed (Participants) | 45 | 37
Percentage of Participants | 80.0 | 78.4
Statistical Analysis 1: Comparison: IMI/REL FDC vs PIP/TAZ FDC; Test type: Other; Adjusted difference in percentage = 1.4, 95% CI 2-sided [-16.5 to 19.8] — Adjusted difference and the 95% CIs are based on Miettinen & Nurminen method stratified by randomization stratum

8. Secondary Outcome: Percentage of Participants Achieving a Favorable Microbiological Response at EOT Visit in the ME Population
Description: Favorable overall microbiological response rates was defined as "eradication" (A lower respiratory tract culture taken at the EOT visit showed eradication of the pathogen found at study entry) OR "presumed eradication" (No specimen taken because participant was deemed clinically cured or improved) of the baseline pathogen. The percentage of participants achieving a favorable microbiological response at End of Treatment (EOT) visit in the ME population is presented.
Time Frame: Up to approximately 14 days
Population: All randomized participants receiving ≥1 dose of IV study therapy without presence of positive cocci (MITT); who met important diagnostic criteria for study with no significant protocol deviation and received minimum duration of IV study therapy (CE); had a baseline bacterial pathogen cause of HABP/VABP against which IMI/REL has antibacterial activity and results from a lower respiratory tract culture obtained at indicated time point (ME); and had non-missing/non-indeterminate response at EOT.
Measure: Number; unit: Percentage of Participants
Arm/Group | IMI/REL FDC | PIP/TAZ FDC
Number analyzed (Participants) | 57 | 47
Percentage of Participants | 71.9 | 74.5
Statistical Analysis 1: Comparison: IMI/REL FDC vs PIP/TAZ FDC; Test type: Other; Adjusted difference in percentage = -3.1, 95% CI 2-sided [-19.8 to 14.4] — Adjusted difference and the 95% CIs are based on Miettinen & Nurminen method stratified by randomization stratum

9. Secondary Outcome: Percentage of Participants Experiencing Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The percentage of participants experiencing an AE was reported for each arm.
Time Frame: Up to approximately 98 days
Population: All randomized participants who received at least 1 dose of IV study therapy were assessed.
Measure: Number; unit: Percentage of Participants
Arm/Group | IMI/REL FDC | PIP/TAZ FDC
Number analyzed (Participants) | 134 | 136
Percentage of Participants | 86.6 | 84.6
Statistical Analysis 1: Comparison: IMI/REL FDC vs PIP/TAZ FDC; Test type: Other; Adjusted difference in percentage = 2.0, 95% CI 2-sided [-6.5 to 10.6] — Difference and the 95% CIs are based on Miettinen & Nurminen method stratified by randomization stratum

10. Secondary Outcome: Percentage of Participants Discontinuing Study Drug Due to AEs
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The percentage of participants that discontinued study therapy due to an AE was reported for each arm.
Time Frame: Up to approximately 14 days
Population: All randomized participants who received at least 1 dose of IV study therapy were assessed.
Measure: Number; unit: Percentage of Participants
Arm/Group | IMI/REL FDC | PIP/TAZ FDC
Number analyzed (Participants) | 134 | 136
Percentage of Participants | 3.7 | 8.1
Statistical Analysis 1: Comparison: IMI/REL FDC vs PIP/TAZ FDC; Test type: Other; Adjusted difference in percentage = -4.4, 95% CI 2-sided [-10.7 to 1.4] — Difference and the 95% CIs are based on Miettinen & Nurminen method stratified by randomization stratum

ADVERSE EVENTS:
Time Frame: Up to approximately 98 days
Description: All-cause mortality: all randomized participants; Safety: all randomized participants who received at least one dose of study treatment.
Groups:
- IMI/REL: Imipenem/cilastatin/relebactam (IMI/REL) was administered intravenously (IV) as a fixed-dose combination (FDC) at a dosage of 500 mg IMI/250 mg REL, once every 6 hours for a minimum 7 days, up to 14 days. At the start of IMI/REL treatment, participants were treated empirically with 600 mg open-label linezolid administered IV every 12 hours until methicillin-resistant Staphylococcus aureus (MRSA) was ruled out. Participants with confirmed MRSA infection continued to receive 600 mg linezolid every 12 hours for a minimum of 7 days, up to 14 days total.
- PIP/TAZ: Piperacillin/tazobactam (PIP/TAZ) was administered IV as a FDC at a dosage of 4000 mg PIP/500 mg TAZ once every 6 hours for a minimum 7 days, up to 14 days. At the start of PIP/TAZ treatment, participants were treated empirically with 600 mg open-label linezolid administered IV every 12 hours until methicillin-resistant Staphylococcus aureus (MRSA) is ruled out. Participants with confirmed MRSA infection continued to receive 600 mg linezolid every 12 hours for a minimum of 7 days, up to 14 days total.
Arm/Group | IMI/REL | PIP/TAZ
All-Cause Mortality (participants affected / at risk) | 18/138 | 11/136
Serious Adverse Events (participants affected / at risk) | 29/134 | 21/136
Other Adverse Events (participants affected / at risk) | 81/134 | 66/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMI/REL (N=134) | PIP/TAZ (N=136)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastropleural fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 2 (2)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Anastomotic fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lung squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 3 (3)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Ruptured cerebral aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 3 (3)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 4 (4) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMI/REL (N=134) | PIP/TAZ (N=136)
Anaemia (Blood and lymphatic system disorders) | 18 (20) | 17 (17)
Constipation (Gastrointestinal disorders) | 15 (15) | 9 (10)
Diarrhoea (Gastrointestinal disorders) | 21 (27) | 22 (25)
Vomiting (Gastrointestinal disorders) | 8 (11) | 6 (6)
Hepatic function abnormal (Hepatobiliary disorders) | 17 (18) | 13 (13)
Urinary tract infection (Infections and infestations) | 8 (8) | 4 (4)
Alanine aminotransferase increased (Investigations) | 12 (12) | 13 (13)
Aspartate aminotransferase increased (Investigations) | 8 (8) | 7 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (14) | 17 (19)
Hyponatraemia (Metabolism and nutrition disorders) | 17 (18) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/33/NCT03583333/Prot_SAP_000.pdf